CLINICAL TRIAL: NCT01896258
Title: A Nationwide Survey of Korean Emergency Department Triage Systems and Scales; a First Step Towards Korean Triage and Acuity Scale(KTAS)
Brief Title: A Nationwide Survey of Korean Emergency Department Triage Systems and Scales
Status: Completed | Type: Observational
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Joonbum Park, M.D., Hanyang University
Other Study IDs: jesumania
Record Dates: First submitted 2013-07-02; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Focus of Study

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Regional emergency centers
- Local emergency centers

SUMMARY:
As a first step towards reform of the emergency medical service system by standardizing triage scale to Korean Triage and Acuity Scale(KTAS), we aimed to assess the present status of our emergency department triage systems and illustrated the present status and problems of the Korean emergency department triage system.

DETAILED DESCRIPTION:
Study design In Korea, EDs are classified into 4 levels, 21 4th degree regional EDs, 115 3rd degree local EDs, 323 2nd degree local emergency facilities and 132 1st degree other emergency facilities. Korea is divided into 21 medical regions according to access to hospitals, the population of cities and their areas. A regional ED is located in each medical region. There is a local ED for every million people in metropolitan areas, and every five hundred thousand peoples in other cities. The investigators selected all 4th and 3rd degree EDs in Korea (21 regional and 115 local EDs; at Dec 31, 2011). The triage systems of these EDs are qualified and controlled by the National Emergency Medicine Center. The investigators conducted a telephone and e-mail survey of triage officers from September 4 to November 27, 2012. The name of each center was identified from the 2011 Annual Report of Korean Emergency Medicine, which included the phone number of each ED.6) Initially, an EM specialist telephoned the nurse manager of all EDs and explained the purpose of the survey. He then selected a triage officer from each ED who had worked in the emergency department for more than 3 years. The interviewer first asked them whether they wanted a telephone interview or the e-mail survey. 102 EDs chose the telephone interview, in which the interviewer read the questions and noted the answers on the survey sheet in a standard order to prevent interviewer bias. The investigators instructed the interviewer not to change the wording or content of any survey question; however if a respondent did not understand the meaning of a word, the interviewer was allowed to explain it. Thirty four EDs wanted to answer by e-mail, and the investigators sent the survey form to them. If the answer did not arrive after a week, the investigators sent the same e-mail again, and after two weeks the investigators called the respondent again. In 4 cases the nurse manager of an ED or the triage officer declined to answer the survey him/herself for security reasons. In those cases, the investigators contacted the hospital administrator and asked him or her to forward an e-mail to the ED triage officer or nurse manager.

Data collection and processing The survey instrument was revised by 6 emergency medicine departments of 2 institutions. (The survey instrument is posted in online as a supplementary file). Data collected included identification of respondents, actual usage of separate triage rooms, occupations of triage officers, presence of documented triage scales, type of triage scale, triage officer's opinion about the problem of his own triage scale, education for the triage officers, and the process of reviewing their triage scales.

The investigators used SPSS 18 (IBM SPSS Inc., Chicago, Illinois, USA) for data management and analysis. The investigators compared characteristics of the regional EDs with those of local EDs and examined aspects of the ED triage systems such as frequency of use of the triage room, occupation of the triage officer and so on. The investigators compared the features of EDs with verified triage scales and those with unverified triage scales, and assessed the quality control of the EDs by asking about education for triage, and verification of the triage scale. This research was reviewed by the University of Hanyang institutional review board and was exempted from written informed consent. Survey respondents were informed that their participation was voluntary and that the results of the survey would be kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* consent to survey

Exclusion Criteria:

* not consent to survey

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: triage officers of 136 emergency centers in Korea
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Emergency departments which have verified triage scales. | Sep, 2012-Nov, 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang university Seoul hospital, Seoul, Seoul, South Korea